CLINICAL TRIAL: NCT06646770
Title: Segmentectomy Versus Lobectomy in Clinical T1c Non-Small Cell Lung Cancer: A Non-Inferiority Trial
Brief Title: SEgmentectomy Versus Lobectomy in T1C Non-Small Cell Lung Cancer (SELTIC)
Acronym: SELTIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Akif Turna, Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2501
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; T1c; Segmentectomy; Lobectomy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Mastectomy, Segmental; Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Segmentectomy (Experimental): Pulmonary anatomic segmentectomy with mediastinal nodal dissection
  Interventions: Procedure: Segmentectomy
- Lobectomy (Active Comparator): Pulmonary lobectomy with mediastinal nodal dissection
  Interventions: Procedure: Lobectomy

INTERVENTIONS:
Procedure: Segmentectomy — Pulmonary anatomic segmentectomy with mediastinal nodal dissection via VATS, RATS or open approach.
  Arms: Segmentectomy
Procedure: Lobectomy — Pulmonary lobectomy with mediastinal nodal dissection via VATS, RATS or open approach.
  Arms: Lobectomy

SUMMARY:
The goal of this clinical trial is to investigate the role of segmentectomy in clinical T1c (2-3 cm) non-small cell lung cancer (NSCLC). The main questions we aim to answer are:

1. Is segmentectomy non-inferior to lobectomy in cT1c NSCLC in terms of overall and recurrence free survival?
2. What are the mortality and morbidity rates of segmentectomy compared to lobectomy?

Researchers will compare segmentectomy and lobectomy in terms of overall and recurrence free survival.

Participants will:

* Undergo either pulmonary lobectomy or segmentectomy with mediastinal nodal dissection
* Be followed up with a chest CT in every 3 months in first year, every 6 months in second year and every year for following 3 years

ELIGIBILITY:
Inclusion Criteria:

* Clinical T1c NSCLC
* Parenchymal nodule >2 cm in diameter
* Parenchymal nodule ≤3 cm in diameter
* Consolidation / Tumor Rate (CTR) ≥ 0.50
* Definitive pathological diagnosis of NSCLC preoperative or intraoperatively
* No evidence of distant metastasis
* No evidence of N2 disease
* Adequate pulmonary functions for lobectomy or segmentectomy

Exclusion Criteria:

* Pure GGO lesions
* Pathologic diagnosis other than NSCLC
* Technically not suitable for simple or complex segmentectomy, or lobectomy
* Evidence of distant metastasis
* Pathologically confirmed N2 or N3 disease
* Major comorbidity that precludes surgery
* Intraoperative mediastinal nodal dissection of less than 3 lymph node stations
* Prior malignancy in five years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Survival Survival | 5 years
  Overall and recurrence free survival

SECONDARY OUTCOMES:
Complication rate associated with surgery | 90 days
Mortality rate | 90 days
  mortality rate associated with surgery

CONTACTS AND LOCATIONS:
Overall Officials: Akif Turna, MD, PhD, Principal Investigator — Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty
Locations (1):
- Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)